CLINICAL TRIAL: NCT05294458
Title: A Single Part, Three-Way Crossover, Randomised, Open-Label Study Designed to Evaluate the Relative and Absolute Bioavailability Following a Single Subcutaneous Injection of a Novel High Concentration Subcutaneous Formulation of Cotadutide Against a Low Concentration Subcutaneous Formulation and Intravenous (IV) Formulation for Reference, in Healthy Subjects
Brief Title: A Randomised, Open-Label Study to Evaluate the Relative and Absolute Bioavailability of Cotadutide in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Quotient Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D5671C00009; 2021-005442-15 (EudraCT Number)
Record Dates: First submitted 2022-03-11; First posted 2022-03-24 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Non-alcoholic Steatohepatitis; Type 2 Diabetes Mellitus (T2DM); Chronic Kidney Disease
Keywords: Steatohepatitis; Diabetes; Kidney disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Diabetes Mellitus, Type 2; Renal Insufficiency, Chronic; Fatty Liver; Diabetes Mellitus; Kidney Diseases | interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cotadutide solution for injection (Experimental): Period 1, subcutaneous injection of cotadutide solution
  Period 2, subcutaneous injection of cotadutide solution
  Period 3, subcutaneous injection of cotadutide solution
  Interventions: Drug: cotadutide solution for injection

INTERVENTIONS:
Drug: cotadutide solution for injection — cotadutide solution for injection

SUMMARY:
The Sponsor is developing the test medicine, cotadutide, for the potential treatment of non-alcoholic steatohepatitis (NASH) and Type 2 Diabetes Mellitus (T2DM) with chronic kidney disease. This healthy volunteer study will try to identify how two different concentrations of cotadutide are taken up by the body when dosed under the skin (subcutaneous injection). The study will also try to identify the absolute bioavailability of cotadutide (amount taken up by the body when dosed under the skin compared to an injection directly into the vein (intravenous)). This is a single-part, three-period study taking place at one non-NHS site in the UK and will involve 12 male and female (non-pregnant/non-lactating) volunteers aged 18-55. For each study period, on Day 1 volunteers will receive cotadutide as either a subcutaneous injection (into the stomach) or an intravenous injection following an overnight fast of at least 10 hours. The subcutaneous injections will be given as either a 1 mg/ml or 5 mg/ml concentration. The intravenous injection will be given as a 0.1 mg/ml concentration. Volunteers will be discharged on Day 4 and there will be a washout period of 7 days between dosing.

Blood samples will be taken at regular intervals for pharmacokinetics and safety assessments from Day -1 to discharge. Volunteers will need to return for a follow up visit 28 (±2) days post-first dose for provisional of an anti-drug antibody sample and to ensure wellbeing

DETAILED DESCRIPTION:
The Sponsor is developing the test medicine, cotadutide, for the potential treatment of non-alcoholic steatohepatitis (NASH) and Type 2 Diabetes Mellitus (T2DM) with chronic kidney disease. NASH is a common liver disease characteristic of a damaged liver that may no longer work properly. T2DM is a condition that causes sugar (glucose) levels in the blood to become too high which can damage the blood vessels within the kidney leading to chronic kidney disease and also causing problems with eyes, heart and nerves. This healthy volunteer study will try to identify how two different concentrations of cotadutide are taken up by the body when dosed under the skin (subcutaneous injection). The study will also try to identify the absolute bioavailability of cotadutide (amount taken up by the body when dosed under the skin compared to an injection directly into the vein (intravenous)). The study will also assess the safety and tolerability of cotadutide.

This is a single-part, three-period study taking place at one non-NHS site in the UK and will involve 12 male and female (non-pregnant/non-lactating) volunteers aged 18-55. For each study period, on Day 1 volunteers will receive cotadutide as either a subcutaneous injection (into the stomach) or an intravenous injection following an overnight fast of at least 10 hours. The subcutaneous injections will be given as either a 1 mg/ml or 5 mg/ml concentration. The intravenous injection will be given as a 0.1 mg/ml concentration. Volunteers will be discharged on Day 4 and there will be a washout period of 7 days between dosing.

Blood samples will be taken at regular intervals for pharmacokinetics and safety assessments from Day -1 to discharge. Volunteers will need to return for a followup visit 28 (±2) days post-first dose for provisional of an anti-drug antibody sample and to ensure wellbeing

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated, written informed consent prior to any study specific procedures.
* Healthy males or non-pregnant, non-lactating healthy females aged 18 to 55 years at the time of signing informed consent.
* Females must have a negative serum pregnancy test at screening and a negative urine pregnancy test on admission to the unit, must not be lactating, confirmed at screening and fulfil the criteria detailed in Section 9.4.
* Have a body mass index (BMI) between 18.0 and 30.0 kg/m2 inclusive and weigh at least 50 kg and no more than 100 kg inclusive.
* Must be willing and able to communicate and participate in the whole study.
* Subjects must have been received both doses of the SARS-CoV-2 vaccine.
* Must agree to adhere to the contraception requirements defined in Section 9.4

Exclusion Criteria:

* History of any clinically significant disease or disorder which, in the opinion of the investigator, may either put the volunteer at risk because of participation in the study, or influence the results or the volunteer's ability to participate in the study.
* History or presence of any disease or condition known to interfere with absorption, distribution, metabolism, or excretion of drugs.
* Evidence of renal impairment at screening, as indicated by an estimated eGFR of <60 mL/min using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation.
* A personal or family history of medullary thyroid carcinoma or have multiple endocrine neoplasia syndrome type 2.
* Thyroid C-cell hyperplasia (calcitonin level > 50 ng/L) or medullary thyroid carcinoma at screening.
* History of clinically significant cardiovascular, renal, hepatic, dermatological, respirator, neurological, psychiatric or gastrointestinal disease disorder including a history of pancreatitis.
* Any clinically significant illness, medical/surgical procedure, or trauma within 4 weeks of the first administration of IMP.
* Any clinically significant abnormalities in clinical chemistry, haematology, or urinalysis results, at screening as judged by the investigator.
* Amylase and/or lipase >1.5 × upper limit of normal (ULN) at screening
* Any clinically significant abnormal findings in vital signs, at screening and/or first admission to the study unit, as judged by the investigator.
* Any clinically significant abnormalities on 12-lead ECG, including but not limited to QTcF >450 msec, at screening, as judged by the investigator.
* Any positive result on screening for serum hepatitis B surface antigen (HBsAg), hepatitis C antibody (HCV Ab), and human immunodeficiency virus (HIV) antibody.
* Evidence of current infection with SARS-Cov-2.
* Has received another new chemical entity (defined as a compound which has not been approved for marketing) within the 90 days prior to Day 1, or less than 5 elimination half-lives prior to Day 1, whichever is longer. Note: subjects consented and screened, but not randomised in this study or a previous phase I study, are not excluded.
* Plasma donation within 1 month of screening or any blood donation/loss more than 500 mL during the 3 months prior to screening.
* History of severe allergy/hypersensitivity or ongoing allergy/hypersensitivity, as judged by the investigator or history of hypersensitivity to drugs with a similar chemical structure or class to cotadutide. Hay fever is allowed unless it is active
* Current smokers or those who have smoked or used nicotine products (including e-cigarettes) within the 3 months prior to screening. A confirmed breath carbon monoxide reading of greater than 10 ppm at screening or admission.
* Positive screen for drugs of abuse at screening or on each admission to the study centre or positive screen for alcohol on each admission to the study centre.
* Use of any prescribed or nonprescribed medication including antacids, analgesics (other than paracetamol/acetaminophen, hormonal contraception and hormonal replacement therapy), herbal remedies, megadose vitamins (intake of 20 to 600 times the recommended daily dose) and minerals during the two weeks prior to the first administration of IMP or longer if the medication has a long half-life. Exceptions may apply, as determined by the investigator, if each of the following criteria are met: medication with a short half-life if the washout is such that no pharmacodynamic activity is expected by the time of dosing with IMP; and if the use of medication does not jeopardize the safety of the trial subject; and if the use of medication is not considered to interfere with the objectives of the study
* Known or suspected history of alcohol or drug abuse in the past 2 years or excessive intake of alcohol (>21 units per week for men and >14 units per week or women [1 unit = ½ pint beer, or a 25 mL shot of 40% spirit, 1.5 to 2 units = 125 mL glass of wine, depending on type]) or as judged by the investigator. A confirmed positive alcohol breath test at screening or admission.
* Excessive intake of caffeine-containing drinks or food (e.g., coffee, tea, chocolate) as judged by the investigator. Excessive intake of caffeine defined as the regular consumption of more than 600 mg of caffeine per day (e.g., >5 cups of coffee) or would likely be unable to refrain from the use of caffeine-containing beverages during confinement at the investigational site.
* Involvement of any Astra Zeneca, Quotient or study site employee or their close relatives.
* Subjects who have previously received cotadutide.
* Any subject who has received a GLP-1 analogue containing preparation within the last 30 days or 5 half-lives of the drug (whichever is longer) at the time of screening.
* Subjects who do not have suitable veins for multiple venepunctures/cannulation as assessed by the investigator or delegate at screening.
* Skin disorder/condition or tattoos in the area of the proposed injection site which can interfere with assessments required by protocol.
* Judgment by the investigator that the volunteer should not participate in the study if they have any ongoing or recent (i.e., during the screening period) minor medical complaints that may interfere with the interpretation of study data or are considered unlikely to comply with study procedures, restrictions, and requirements.
* Subjects who cannot communicate reliably with the investigator.
* Vulnerable subjects, e.g., kept in detention, protected adults under guardianship, trusteeship, or committed to an institution by governmental or juridical order.
* Failure to satisfy the investigator of fitness to participate for any other reason.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2022-03-28 (Actual); Primary Completion 2022-09-12 (Actual); Study Completion 2022-09-12 (Actual)

PRIMARY OUTCOMES:
Absolute bioavailability of the high and the low concentration cotadutide SC formulations | Collection of plasma samples from pre-dose to 72 hours post-dose.
  Evaluation of the absolute bioavailability (F) of the SC formulations by comparison of AUCsubcut/AUCIV
Maximum observed concentration (cmax) | Collection of plasma samples from pre-dose to 72 hours post-dose.
  Assessment of pharmacokinetics and relative bioavailability of cotadutide solution for injection by measuring maximum observed concentration (cmax)
Relative bioavailability of a high concentration cotadutide SC formulation in comparison to low concentration formulation, in the fasted state | Collection of plasma samples from pre-dose to 72 hours post-dose.
  Pharmacokinetic parameters AUC0-t for cotadutide in the high concentration and low concentration regimens
Relative bioavailability of a high concentration cotadutide SC formulation in comparison to low concentration formulation, in the fasted state | Collection of plasma samples from pre-dose to 72 hours post-dose.
  Pharmacokinetic parameters AUC0-inf for cotadutide in the high concentration and low concentration regimens

SECONDARY OUTCOMES:
Provide additional details on the single dose PK of cotadutide | Collection of plasma samples from pre-dose to 72 hours post-dose.
  Pharmacokinetic parameters tmax, for cotadutide, as applicable
Provide additional details on the single dose PK of cotadutide | Collection of plasma samples from pre-dose to 72 hours post-dose.
  Pharmacokinetic parameters Cmax, for cotadutide, as applicable
Provide additional details on the single dose PK of cotadutide | Collection of plasma samples from pre-dose to 72 hours post-dose.
  Pharmacokinetic parameters AUC0-t, for cotadutide, as applicable
Provide additional details on the single dose PK of cotadutide | Collection of plasma samples from pre-dose to 72 hours post-dose.
  Pharmacokinetic parameters AUC0-inf, for cotadutide, as applicable
Provide additional details on the single dose PK of cotadutide | Collection of plasma samples from pre-dose to 72 hours post-dose.
  Pharmacokinetic parameters t1/2, for cotadutide, as applicable
Provide additional details on the single dose PK of cotadutide | Collection of plasma samples from pre-dose to 72 hours post-dose.
  Pharmacokinetic parameters λz, for cotadutide, as applicable
Provide additional details on the single dose PK of cotadutide | Collection of plasma samples from pre-dose to 72 hours post-dose.
  Pharmacokinetic parameters CL (IV dose), for cotadutide, as applicable
Provide additional details on the single dose PK of cotadutide | Collection of plasma samples from pre-dose to 72 hours post-dose.
  Pharmacokinetic parameters CL/F, for cotadutide, as applicable
Provide additional details on the single dose PK of cotadutide | Collection of plasma samples from pre-dose to 72 hours post-dose.
  Pharmacokinetic parameters Vz, for cotadutide, as applicable
Provide additional details on the single dose PK of cotadutide | Collection of plasma samples from pre-dose to 72 hours post-dose.
  Pharmacokinetic parameters Vz/F, for cotadutide, as applicable
Provide additional details on the single dose PK of cotadutide | Collection of plasma samples from pre-dose to 72 hours post-dose.
  Pharmacokinetic parameters MRTinf, for cotadutide, as applicable
Number of adverse events (AEs) experienced by subjects | Collection of plasma samples from pre-dose to 72 hours post-dose.
  Safety and tolerability assessed through the incidence of AEs
Evaluate immunogenicity for cotadutide administered as low and high concentration SC formulations and an IV formulation | Collection of plasma samples from pre-dose to 72 hours post-dose.
  ADA incidence and titre

OTHER OUTCOMES:
To collect data on the size and shape of SC injection | before and immediately after injection and up to 72 hours post-injection
  Measurement of thermal image of the injection point before and immediately after injection and up to 72 hours post-injection
Temperature needed at the injection site to homogenize at the point of injection | Before and immediately after injection and up to 72 hours post-injection
  Measurement of thermal image of the injection point before and immediately after injection and up to 72 hours post-injection

CONTACTS AND LOCATIONS:
Overall Officials: Somasekhara Menakuru, MBBS, MS, MRCS, DPM, MFPM, Principal Investigator — Quotient Sciences
Locations (1):
- Research Site, Ruddington, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: The redacted CSR D5671C00009 — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5671C00009&attachmentIdentifier=30a648c8-396e-40e9-b1d2-6e99994abd37&fileName=The_redacted_CSR_D5671C00009.pdf&versionIdentifier=